CLINICAL TRIAL: NCT00665730
Title: Evaluation of the Safety and Effectiveness of Sepraspray™ in Limiting the Formation of Postoperative Adhesions to Serosal Tissue (Abdominal Surgery)
Brief Title: Evaluation of the Safety and Effectiveness of Sepraspray™ in Reducing Post-surgical Adhesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to low enrollment.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SSPRAY00406
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Abdominal Adhesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sepraspray (Experimental): Sepraspray Powder applied on the viscera directly under the midline incision followed by incision closure. Sepraspray dose applied was between 2 g and 4 g per patient.
  Interventions: Device: Sepraspray
- Control (No Intervention): No anti-adhesion treatment used.

INTERVENTIONS:
Device: Sepraspray
  Arms: Sepraspray

SUMMARY:
This study will examine the safety and efficacy of Sepraspray in the following model of abdominal surgery: total proctocolectomy and pelvic pouch with diverting ileostomy via laparotomy to treat ulcerative colitis or familial polyposis. Adhesion formation will be evaluated laparoscopically at ileostomy take down. NOTE: A decision was made to terminate this study in June 2008 due to low enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo a total proctocolectomy and a pelvic pouch with diverting ileostomy.

Exclusion Criteria:

* Patients who are pregnant.
* Patients with ongoing abdominal abscess.
* Patients with ongoing bacterial peritonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Efficacy: Primary efficacy endpoints include the incidence of adhesions to the midline incision | 8-14 weeks

SECONDARY OUTCOMES:
Secondary: efficacy endpoints include the extent of adhesions to the midline incision and the severity of adhesions to the midline incision. | 8-14 weeks
Safety: safety endpoints include assessments of adverse events, vital signs, incisional wound healing, clinical laboratory evaluations, and concomitant medications. | 8-14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (6):
- Czechia (2):
  - Masarykova
  - Prague
- Aarhus C, Denmark
- Lille, France
- Heidelberg, Germany
- Cottingham, East Yorkshire, United Kingdom